CLINICAL TRIAL: NCT06983626
Title: Predictive Factors of Successful Micro-dissection Testicular Sperm Extraction For Patients With Non Obstructive Azoospermia
Brief Title: Management of Non Obstructive Azoospermia in Men
Acronym: azoospermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Hafez Badawy Hafez, assistant lecturer of urology, South Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SVU MED URO016 2 22 5 401
Record Dates: First submitted 2025-04-28; First posted 2025-05-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Male Infertility; Azoospermia, Nonobstructive
MeSH Terms: conditions — Infertility, Male; Azoospermia, Nonobstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- male infertility (Active Comparator): azoospermia non obstructive type
  Interventions: Procedure: micro-dissection testicular sperm extraction

INTERVENTIONS:
Procedure: micro-dissection testicular sperm extraction — dissection of the seminefrous tubules under microscope to extract sperms
  Other Names: TESE; TESA; PESA

SUMMARY:
this study predicts the factors of successful micro testicular sperm extraction in azoospermia patients in male infertility

DETAILED DESCRIPTION:
primary outcomes: these factors were the age, testicular size, hormonal, evidence of varicocles and the out come of Micro_TESE secondary outcomes: make good decision for Micro-TESE with low economic laboratory and radiology requirement As every failed microTESE-ICSI procedure exposes the couple to an emotional, financial burden and increase the incidence of complication such as bleeding, hematoma and testicular atrophy

ELIGIBILITY:
Inclusion Criteria: Non obstructive Azoospermia with no genetic abnormalties as klinefelter syndrome

* redo Micro TESE

Exclusion Criteria:

* obstructive Azoospermia and bilateral congenital absent of vas

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Sperm Retrieval Success Rate and identification of Predictive Factors | 1st 1 year
  Determine which preoperative factors are significantly associated with successful sperm retrieval. These may include:
  Serum Follicle-Stimulating Hormone (FSH) Levels: Elevated FSH levels have been linked to reduced sperm retrieval success.
  And patient Age and testicular size to reach the best one to predict the success rate

SECONDARY OUTCOMES:
Assess the success rates of ART procedures following sperm retrieval and complications | 2 years
  Assisted Reproductive Technology (ART) Outcomes
  Fertilization Rates: The percentage of oocytes successfully fertilized.
  Embryo Development: Quality and progression of embryos to the blastocyst stage.
  Clinical Pregnancy Rates: Confirmed pregnancies via ultrasound.
  Live Birth Rates: The ultimate success metric of ART procedures
  Complication Rates
  Monitor and document any complications arising from the sperm retrieval procedure, such as:
  Testicular Hematoma
  Infection
  Testicular Atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Gamal abdelhammid alsagheer, professour of urology, professour, Study Director — South Valley University
Locations (1):
- Faculty of Medicine, South Valley University, Luxor, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
according to the results
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: urologist and andrologist
URL: https://svuijm.journals.ekb.eg/

REFERENCES:
- See also: Azoospermia — https://pubmed.ncbi.nlm.nih.gov/32519242/